CLINICAL TRIAL: NCT00935402
Title: Sleep Deprivation and Energy Balance
Acronym: Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Clinilabs, Inc. (Other); Columbia University (Other)
Responsible Party: Marie-Pierre St-Onge/Research Associate, St. Luke's/Roosevelt Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01HL091352-01A1 (NIH); R01HL091352-01A1 (NIH)
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-05

CONDITIONS: Obesity
Keywords: Energy balance; Weight management; Food intake; Energy expenditure
MeSH Terms: conditions — Obesity | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Sleep (Experimental): Subjects are permitted to spend 4 hours in bed per night for 5 consecutive nights. Subjects are inpatients for a period of 6 days.
  Interventions: Behavioral: Sleep
- Regular Sleep (Active Comparator): Subjects are permitted to spend 9 hours in bed per night for 5 nights. Subjects are inpatients for a period of 6 days.
  Interventions: Behavioral: Sleep

INTERVENTIONS:
Behavioral: Sleep — Subjects are randomly assigned to one of 2 arms sequence: short followed by regular or regular followed by short. Each arm is 6 days in length and separated by a 2-4 week washout period.

SUMMARY:
Observational and epidemiological studies have found a link between obesity and short sleep duration with the prevalence of both increasing in the past decades. At this time, it is unknown whether short sleep is a cause of obesity and how short sleep would lead to obesity. Some studies associate short sleep with increased levels of hormone that stimulate appetite. This study will examine how food intake and energy expenditure can be modified by sleep duration as a means of understanding a potential causal pathway.

DETAILED DESCRIPTION:
Recent epidemiological studies show that short sleep duration (≤5-7 h/night) correlates with overweight and obesity, such that individuals with short sleep periods tend to have a higher body mass index (BMI) than those who sleep 8-9 h/night. The mechanism for this relationship is currently unknown. However, energy balance must be disrupted to produce weight gain. Therefore, the purpose of this study is to examine the impact of short sleep duration, 4 h/night, relative to habitual sleep duration of 8-9 h/night, on energy balance. The major aims of this study are to compare energy expenditure and energy intake during the periods of habitual and short sleep duration and to examine the neural and hormonal pathways involved in eating behavior under periods of habitual and short sleep. Men and women, 30-45 y and BMI 22-25 kg/m2, will be recruited to participate in this randomized, crossover study of short and habitual sleep periods. During each period of 5 nights, subjects will be required to sleep at the laboratory under supervision. During this time, subjects will be total inpatients to ensure compliance with the protocol. Each sleep duration period will be separated by a 2-4-wk washout period. On the first day of each phase, subjects will be given a dose of doubly-labeled water to measure free-living energy expenditure over the 6-d period. During the first 4 days, energy intake will be controlled and meals served at fixed times. The last 2 days will be ad libitum feeding of self-selected meals. Hormones, including leptin, insulin, ghrelin, PYY, adiponectin, and GLP-1 will be assessed daily in the fasted state and, on day 4, over a 24-hour period, while subjects are consuming a controlled diet with fixed meal times. Functional magnetic resonance imaging measurements of brain activity in response to food stimuli will be done on day 5 to examine brain regions associated with motivation to eat. On day 5, subjects will undergo measurements of basal metabolic rate using indirect calorimetry. Ad libitum energy intakes will be assessed on days 5 and 6. Polysomnographic monitoring will be performed nightly to assess sleep duration. Mediation analyses will allow us to determine whether hormone levels are related to and predictive of energy expenditure and energy intake data. The measurements performed in this study will allow us to determine how reduced sleep periods can impact energy balance and potentially lead to changes in body weight. As such, it will provide comprehensive information of the neural, physiological, hormonal, and behavioral networks related to energy balance and which are affected by sleep duration.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 22-25 kg/m2
* Right-handed
* Sleep 7-9 hours/night
* Normal score on Pittsburgh Quality of Sleep questionnaire, Epworth Sleepiness Scale, Berlin Questionnaire, Sleep Disorders Inventory Questionnaire, Beck Depression Inventory, Composite Scale of Morningness/Eveningness

Exclusion Criteria:

* Smoker
* Neurological, medical, or psychiatric disorder
* Diabetics
* History of eating disorders
* Sleep disorders
* Travel across time zones within 4 weeks of the study
* History of drug and alcohol abuse
* Shift worker
* Caffeine intake > 300 mg/d
* Excessive daytime sleepiness
* Regular napping
* History of drowsy driving
* Pregnancy or within 1 y post-partum
* Heavy equipment operator or commercial long-distance driver
* Contra-indications for MRI scanning

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate | Day 5 of each arm
Food intake | Days 5-6 of each arm
Hormone Measurements | Daily fasting, and every 2 hours on day 4 of each arm
Regional brain activity | Day 6 of each arm
Energy expenditure | Each 6 day arm

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Ph.D, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (3):
- United States (3):
  - Clinilabs, New York, New York
  - St. Luke's/Roosevelt Hospital, New York, New York
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Smith I, Salazar I, RoyChoudhury A, St-Onge MP. Sleep restriction and testosterone concentrations in young healthy males: randomized controlled studies of acute and chronic short sleep. Sleep Health. 2019 Dec;5(6):580-586. doi: 10.1016/j.sleh.2019.07.003. Epub 2019 Aug 12. PMID 31416797
- [Derived] McNeil J, St-Onge MP. Increased energy intake following sleep restriction in men and women: A one-size-fits-all conclusion? Obesity (Silver Spring). 2017 Jun;25(6):989-992. doi: 10.1002/oby.21831. Epub 2017 Apr 12. PMID 28401667
- [Derived] St-Onge MP, Roberts A, Shechter A, Choudhury AR. Fiber and Saturated Fat Are Associated with Sleep Arousals and Slow Wave Sleep. J Clin Sleep Med. 2016 Jan;12(1):19-24. doi: 10.5664/jcsm.5384. PMID 26156950
- [Derived] Shechter A, St-Onge MP. Delayed sleep timing is associated with low levels of free-living physical activity in normal sleeping adults. Sleep Med. 2014 Dec;15(12):1586-9. doi: 10.1016/j.sleep.2014.07.010. Epub 2014 Sep 2. PMID 25311835
- [Derived] St-Onge MP, Wolfe S, Sy M, Shechter A, Hirsch J. Sleep restriction increases the neuronal response to unhealthy food in normal-weight individuals. Int J Obes (Lond). 2014 Mar;38(3):411-6. doi: 10.1038/ijo.2013.114. Epub 2013 Jun 19. PMID 23779051
- [Derived] St-Onge MP, O'Keeffe M, Roberts AL, RoyChoudhury A, Laferrere B. Short sleep duration, glucose dysregulation and hormonal regulation of appetite in men and women. Sleep. 2012 Nov 1;35(11):1503-10. doi: 10.5665/sleep.2198. PMID 23115399
- [Derived] St-Onge MP, McReynolds A, Trivedi ZB, Roberts AL, Sy M, Hirsch J. Sleep restriction leads to increased activation of brain regions sensitive to food stimuli. Am J Clin Nutr. 2012 Apr;95(4):818-24. doi: 10.3945/ajcn.111.027383. Epub 2012 Feb 22. PMID 22357722
- [Derived] St-Onge MP, Roberts AL, Chen J, Kelleman M, O'Keeffe M, RoyChoudhury A, Jones PJ. Short sleep duration increases energy intakes but does not change energy expenditure in normal-weight individuals. Am J Clin Nutr. 2011 Aug;94(2):410-6. doi: 10.3945/ajcn.111.013904. Epub 2011 Jun 29. PMID 21715510